CLINICAL TRIAL: NCT06175793
Title: ASPIRE: Adapting Self-Blood Pressure Monitoring to Reduce Health Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00104818; 22.075E (Other: Advocate HC IRB)
Record Dates: First submitted 2023-12-01; First posted 2023-12-19 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASPIRE Intervention Arm (Experimental): The intervention arm will receive usual care, a free blood pressure cuff in addition to the ASPIRE Components.
  Interventions: Behavioral: ASPIRE Intervention
- Control Arm (No Intervention): The control group will receive usual care and a free blood pressure cuff.

INTERVENTIONS:
Behavioral: ASPIRE Intervention — In addition to usual care and a free blood pressure cuff, participants in the intervention arm will receive the ASPIRE components: (1) ASPIRE Tool Kit, (2) ASPIRE Coach, (3) SMBP EHR Documentation, and (4) screening and addressing SDOHs.
  Arms: ASPIRE Intervention Arm

SUMMARY:
The goal of this study is to implement a pilot focusing on developing training manuals and materials for patients and the clinical team to ensure our intervention is delivered consistently and systematically for each patient.

DETAILED DESCRIPTION:
Barriers to blood pressure control are multi-faceted and a silver-bullet solution/intervention does not exist. Therefore, the literature highlights the importance of creating multi-component interventions when addressing blood pressure control. The ASPIRE intervention consists of 5 components identified based on the study team's prior work and review of the literature.

Patients randomized to the intervention arm will receive all 5 components of the ASPIRE intervention. Patients randomized to the control arm will receive only the first component of the ASPIRE intervention and will continue to receive usual care. The ASPIRE intervention consists of 5 components aimed at supporting both patients and clinic care teams in successfully adopting self-measured blood pressure (SMBP) into their clinic workflow.

The 5 ASPIRE components are:

1. Access to cuff (Patient). Patients in the intervention arm and control arm will be measured for and will receive a blood pressure monitoring device to take home and keep beyond the study timeline.
2. Training (Patient). Only patients in the intervention arm will receive training and support on how to accurately measure their blood pressure. They will receive a folder containing an infographic that demonstrates how to accurately measure blood pressure at home. They will also receive a lifestyle infographic describing what they can do to improve their blood pressure.
3. Clear instructions (Patient). Patients in the intervention arm will also receive clear instructions on how to keep a record of their home blood pressure measures and share with their care team. They will be provided with a 7-day blood pressure long that details the number of blood pressure values they need to take in the mornings and evenings for seven days. Additionally, a clinic care team member serving as the ASPIRE coach will follow up with the intervention patients via a scheduled virtual call one week after they receive their materials (blood pressure monitoring device, infographics, and 7-day blood pressure log) to provide further support and instructions on self-measured blood pressure and to emphasize the importance of returning the blood pressure values to their care team.
4. SMBP EHR Documentation (ASPIRE Coach). To facilitate documentation of home blood pressure values in the electronic health record (EHR), the ASPIRE coach will average the blood pressure values patients return and document that average in the EHR. These home blood pressure averages will be shared with the patient's doctor who can use these values to modify treatment as appropriate.
5. Address Social Determinants of Health (Patient). Patients will be screened for social needs via a social determinants of health (SDOH) questionnaire that they will be asked to return to the care team. During the one week follow up virtual call the ASPIRE coach will address any identified social needs by following up with referrals as needed.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Adults >=18 years old
* At least a 1-year history of hypertension
* Must have at least one clinic visit during the study recruitment period (qualifying visit)
* An elevated blood pressure value during their qualifying visit (defined as SBP above 140mm/Hg or DBP above 90mm/Hg)
* Must be on at least one blood pressure lowering medication
* Able to provide consent

Exclusion Criteria:

* Patients residing in a nursing home or receiving home health care
* Patients that don't speak English

Providers:

Inclusion Criteria: Care team members who participate in the study clinic.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
SMBP Feasibility | 1 month
  Feasibility of study methods will be evaluated using EHR data and returned SMBP logs and will include recruitment rates following patient's hypertension visits and loss to follow up rate over the 1 month follow up period.

SECONDARY OUTCOMES:
Change in systolic blood pressure (SBP) | 3 months
  difference in the mean change in SBP (mmHg) between the intervention and control arms
Change in diastolic blood pressure (DBP) | 3 months
  difference in the mean change in DBP (mmHg) between the intervention and control arms
Blood pressure control | 3 months
  proportion of patients with controlled blood pressure (mmHg)
Medication intensification | 3 months
  proportion of patients who had a medication intensification.

OTHER OUTCOMES:
Patient and Care Team Acceptability | 1 month
  Patient and care team acceptability of the research methods and ASPIRE components will be evaluated based on in-depth interviews.
Patients and Care Team Satisfaction | 1 month
  Patient and care team satisfaction with the research methods and ASPIRE components will be evaluated based on in-depth interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Khatib, PhD, Principal Investigator — Advocate Aurora Research Institute
Locations (1):
- ADMG Oak Lawn IM Clinci, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khatib R, Glowacki N, Guzman I, Ozoani O, Brill J, Lauffenburger JC, Biskis A, Gordon M. Adopting Self-Measured Blood Pressure Monitoring Among Underserved Communities (ASPIRE): A Pilot Randomized Controlled Trial. J Gen Intern Med. 2025 Dec;40(16):3822-3830. doi: 10.1007/s11606-025-09646-9. Epub 2025 Jun 25. PMID 40562882
- [Derived] Khatib R, Glowacki N, Guzman I, Shields M, Chase J, Gordon M. Adapting self-measured blood pressure monitoring to reduce health disparities (ASPIRE): a pilot hybrid effectiveness-implementation study protocol. Pilot Feasibility Stud. 2025 Jan 15;11(1):7. doi: 10.1186/s40814-024-01588-z. PMID 39815379